CLINICAL TRIAL: NCT03432975
Title: Evaluation of Multiple Subgingival Irrigations With 10% Povidone Iodine After Scaling and Root Planing : a Randomized Clinical Trial
Brief Title: Evaluation of Multiple Subgingival Irrigations.
Acronym: POLYVIDONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/06NOV/503
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Periodontitis, Adult
MeSH Terms: conditions — Chronic Periodontitis | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: 20 patients (=40 half-mouth); 20 half-mouth per group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Povidone Iodine 10% (Experimental): The side of the mouth receiving the subgingival irrigations of povidone iodine.
  Interventions: Drug: Povidone-Iodine 10%
- Sterile saline solution (Placebo Comparator): The other side of the mouth will be irrigated with a sterile saline solution.
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Povidone-Iodine 10% — The side of the mouth receiving the subgingival irrigations of povidone iodine 10% (test group)
  Arms: Povidone Iodine 10%
Drug: Saline Solution — The other side of the mouth will be irrigated with a sterile saline solution (control group)
  Arms: Sterile saline solution

SUMMARY:
The study will be conducted at the Department of Periodontology, Cliniques universitaires Saint Luc. Patients diagnosed with Generalized Chronic Periodontitis (GChP) based on the current classification of the American Academy of Periodontology will be included. Detailed medical, periodontal and dental history will be obtained. Those who will fulfill the inclusion/exclusion criteria will be invited to participate in the study.

DETAILED DESCRIPTION:
The study will be conducted at the Department of Periodontology, Cliniques universitaires Saint Luc. The patients will be informed in detail of the nature and course of study, and will sign informed consent prior to engagement in the study. Patients diagnosed with GChP based on the current classification of the American Academy of Periodontology will be included. Detailed medical, periodontal and dental history will be obtained. Those who will fulfill the inclusion/exclusion criteria will be invited to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 30 years of age
* At least 15 teeth (excluding third molars and teeth with advanced decay indicated for extraction)
* Any history of periodontal treatment in the previous 6 months
* No removable prosthesis
* A minimum of 6 teeth with at least one site each with periodontal probing depth (PPD) and clinical attachment level (CAL) ≥5 mm
* At least 30% of the sites with PPD and CAL ≥4 mm and bleeding on probing (BOP)

Exclusion Criteria:

* Any sensitivity or allergy to any of the products that will be used in the study
* Thyroid dysfunction
* Systemic disease (ASA II or more)
* Need for antibiotic pre-medication for routine dental therapy
* Antibiotic therapy in the previous 3 months
* Pregnancy and breastfeeding
* Current smokers (more than 5 cigarettes a day)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects reaching ≤ 4 mm in periodontal sites with PPD ≥ 5 mm | up to 6 months
  The primary objective of this study is to determine the effect of PVI on periodontal probing depth (PPD).

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium